CLINICAL TRIAL: NCT01624779
Title: The Effect of Intrathecal Transplantation of Autologous Adipose Tissue Derived Mesenchymal Stem Cells in the Patients With Spinal Cord Injury, Phase I Clinical Study
Brief Title: Intrathecal Transplantation Of Autologous Adipose Tissue Derived MSC in the Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KOR-01
Record Dates: First submitted 2012-06-18; First posted 2012-06-21 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Cord Injury
Keywords: autologous adipose tissue
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: autologous adipose tissue derived mesenchymal stem cells — autologous adipose tissue derived mesenchymal stem cells 9x107cells / 3mL Day 1 and Month 1&2

SUMMARY:
The effect of intrathecal transplantation of autologous adipose tissue derived mesenchymal stem cells in the patients with spinal cord injury, Phase I Clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who don't have any possiblity of improving neurological function despite performed the optimal treatment after spinal cord injury
2. No change in neurological function for 4weeks interval by at least 2 clincal medical specialists
3. Patient who is able to give written informed consent of clinical trial about stemcells treatment

Exclusion Criteria:

1. Patient who is under 19 years and over 70years
2. Patient who must use the mechanical ventilator
3. Patient who have a history of malignant tumor within 5 years
4. Patient who is having a infectious disease of including current hepatitis and HIV
5. Patient who had the brain or spinal cord injury before the spinal cord injury (confirm subject's history from their medical history)
6. Patient who is having a acute disease judged by principle investigator or having a fever over 38.0 ℃ at the vaccination day
7. Patient who is having an anemia or thrombopenia
8. Patient who is having an angina, myocardial infarct, myocardiopathy, obstructive vessel disease, chronic renal failure, glomerulopathy and chronic obstruent lung disease (confirm subject's history from their medical history)
9. Patient who is having a Congenital Immune Deficiency Syndrome or AIDS (confirm subject's history from their medical history)
10. Patient who is having an amyotrophia or joint atrophy
11. Patient who is having an disturbanace of consciousness or dysphrasia
12. Patient who is taking an immunosuppressive agents or corticosteroids agents or cytotoxic agents or needed administration
13. Patient who have experienced another clinical trials within 3 months involving this clinical trial
14. Patient who can't participate in this clinical trial having any opinion regarded as clinical significance judged by principle investigator

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Significant MRI Change before and after intervention | 6 month

SECONDARY OUTCOMES:
Significant neurologic funtion Change before and after intervention | 6 month
Significant Electrophysiological Change before and after intervention | 6 month
Adverse event | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Taehyeong Jo, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbukgu, South Korea